CLINICAL TRIAL: NCT01200082
Title: Sulfation of Bile Acids as a Biomarker for Hepatobiliary Diseases
Status: Terminated | Type: Observational
Why Stopped: Institutional Review Board approval not maintained
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0487-10-EP
Record Dates: First submitted 2010-08-31; First posted 2010-09-13 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Hepatobiliary Diseases
Keywords: chronic hepatitis C/B; alcoholic liver disease; primary biliary cirrhosis; primary sclerosing cholangitis; progressive familial intrahepatic cholestasis
MeSH Terms: conditions — Digestive System Diseases; Liver Diseases, Alcoholic; Liver Cirrhosis, Biliary; Cholangitis, Sclerosing; Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from healthy volunteers at their 1st visit. Urine samples will be obtained from healthy controntrols and patients with hepatobiliary diseases over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Male or female, age 19-65, no apparent signs of hepatobiliary diseases
- Patients with hepatobiliary diseases: Male or female, age 19-65, visiting the UNMC hepatology clinic for treatment from hepatobiliary diseases

SUMMARY:
The investigators hypothesize that the extent of sulfation of toxic BAs and their urinary elimination can be used as a biomarker to predict the severity and prognosis of hepatobiliary diseases. The investigators rationale in this project is that the discovery of biomarkers specific to liver injury would provide the foundation for a specific and non-invasive tool to evaluate disease prognosis, determine patients with higher risk of developing end-stage liver diseases, and determine patients with higher risk of recurrence of hepatobiliary complications after liver transplant.

Patients on the liver transplant list are continuously monitored during their hospitalization and are scheduled for follow-up visits for 12 months after their release post-surgery. Disease progression will be evaluated by monitoring MELD scores, survival, incidence of liver transplant, and incidence of complications related to hepatobiliary conditions such as fluid retention, GI bleeding, encephalopathy, and biliary stricture complications.

DETAILED DESCRIPTION:
The investigators propose the following specific aims to test the investigators hypothesis:

Specific Aim #1: Establish a baseline of individual and total urinary BAs and BA-sulfates in healthy controls and patients with hepatobiliary diseases. A baseline reference of the average and distribution of the percentage of urinary BA-sulfates will be determined in healthy subjects and in patients with hepatobiliary diseases including chronic hepatitis C/B, alcoholic liver disease, hereditary, drug-induced, and autoimmune hepatobiliary diseases. The investigators working hypothesis is that patients' capability to sulfate total or specific BAs, as determined by the percentage of total or specific BAs excreted in the sulfate form, can predict the severity of hepatobiliary diseases, as determined by mayo model for end-stage liver disease (MELD) score and compensation status(compensated and decompensated). Patients with higher MELD score are considered to be at higher risk of developing severe hepatobiliary complications.

Specific Aim #2: Determine the relationship between BA sulfation and the progression of hepatobiliary diseases. This is an exploratory aim to collect preliminary data on the relationship between urinary BAs and the progression of hepatobiliary diseases in liver-transplant and non-liver-transplant patients, as monitored over a1-year period. The investigators working hypothesis is that patients' capabilities of sulfating BAs determine the progression of the disease.

ELIGIBILITY:
Healthy Controls

Inclusion Criteria:

* Male or female, age 19-65, no apparent signs of hepatobiliary diseases

Exclusion Criteria:

* Levels higher than 50, 56, 78 U/L for ALT, AST, and GGT, respectively.

Patient Population

Inclusion Criteria:

* Male or female, age 19-65, visiting the UNMC hepatology clinic for treatment from hepatobiliary diseases

Exclusion Criteria:

* MELD score less than 6

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls: Subjects with no apparemt hepatobiliary diseases Patient Populaton: Subjects visiting the hepatology clinic in UNMC as part of their treatment of hepatobiliry diseases
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Urinary bile acid indexes | Healthy controls: 4 visits over 28 days. Patients: urine collction at every visit as decided in their course of treatment
  Bile acids (BAs), the end products of cholesterol metabolism, are synthesized in liver and excreted into bile, which flows to the small intestine via the bile duct. Most of the BAs are reabsorbed from the intestine into the portal circulation and undergo enterohepatic recirculation with minimal levels detected in urine and blood under normal conditions.

SECONDARY OUTCOMES:
mayo model for end-stage liver disease score (MELD) | Healthy controls: 1st visit only (1 week). Patients: every time a MELD score is required by hepatologists as partrt of their regular course of treatment (1 year)
  MELD score= 3.8*loge (bilirubin [mg/dL]) + 11.2*loge (INR) + 9.6*loge (creatinine [mg/dL]).

CONTACTS AND LOCATIONS:
Overall Officials: Yazen M Alnouti, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medial Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Simko V, Michael S. Urinary bile acids in population screening for inapparent liver disease. Hepatogastroenterology. 1998 Sep-Oct;45(23):1706-14. PMID 9840133
- [Background] Makino I, Hashimoto H, Shinozaki K, Yoshino K, Nakagawa S. Sulfated and nonsulfated bile acids in urine, serum, and bile of patients with hepatobiliary diseases. Gastroenterology. 1975 Mar;68(3):545-53. PMID 1112456
- [Background] Alme B, Bremmelgaard A, Sjovall J, Thomassen P. Analysis of metabolic profiles of bile acids in urine using a lipophilic anion exchanger and computerized gas-liquid chromatorgaphy-mass spectrometry. J Lipid Res. 1977 May;18(3):339-62. PMID 864325